CLINICAL TRIAL: NCT00787202
Title: A Randomized, Placebo Controlled, Double Blind, Parallel Group Multi-Center Study In Order To Investigate Safety And Efficacy Of CP- 690 550 In Subjects With Moderate To Severe Ulcerative Colitis.
Brief Title: A Study To Investigate The Safety And Efficacy Of CP- 690,550 In Patients With Moderate And Severe Ulcerative Colitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921063
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-03

CONDITIONS: Ulcerative Colitis
Keywords: treatment of ulcerative colitis; CP 690 550
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 15 mg BID (Experimental)
  Interventions: Drug: CP- 690 550
- 10 mg BID (Experimental)
  Interventions: Drug: CP- 690 550
- 3 mg BID (Experimental)
  Interventions: Drug: CP- 690 550
- 0.5 mg BID (Experimental)
  Interventions: Drug: CP- 690 550
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: CP- 690 550 — Administration via oral route twice daily for the duration of treatment
  Arms: 15 mg BID
Drug: CP- 690 550 — Administration via oral route twice daily for the duration of treatment
  Arms: 10 mg BID
Drug: CP- 690 550 — Administration via oral route twice daily for the duration of treatment
  Arms: 3 mg BID
Drug: CP- 690 550 — Administration via oral route twice daily for the duration of treatment
  Arms: 0.5 mg BID
Other: placebo — Administration via oral route twice daily for the duration of treatment
  Arms: Placebo

SUMMARY:
The hypothesis of the study is that at least one dose of CP 690 550 is superior to placebo (inactive drug) in inducing remission in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age at screening
* Males and female patients with clinical diagnosis of ulcerative colitis ≥3 months prior to entry into the study.
* Male and female patients with active currently moderate to severe ulcerative colitis defined by Mayo score of ≥6
* Patients with endoscopic sub-score of ≥2 on the Mayo score determined within 7 days of baseline.

Exclusion Criteria:

* Diagnosis of Crohn's disease or diagnosis of indeterminate colitis
* Treatment naive subjects who have not had previous exposure to treatment for ulcerative colitis
* Patients that are currently receiving immunosuppressants, anti-TNFα therapy or interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (56):
- Belgium (3):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Chile (3):
  - Pfizer Investigational Site, Independencia, Santiago Metropolitan
  - Pfizer Investigational Site, Independencia, Santiago RM
  - Pfizer Investigational Site, Viña del Mar
- Czechia (4):
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Usti N. Labem
  - Pfizer Investigational Site, Ústí nad Labem
- Denmark (2):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Aarhus C
- France (4):
  - Pfizer Investigational Site, Lille, France
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Nantes
- Hungary (11):
  - Pfizer Investigational Site, Békéscsaba
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Győr
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Kaposvár
  - Pfizer Investigational Site, Miskolc
  - Pfizer Investigational Site, Mosonmagyaróvár
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szekszárd
  - Pfizer Investigational Site, Szentes
- Israel (3):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Roma
- Mexico (2):
  - Pfizer Investigational Site, Delegacion Benito Juarez, Mexico DF
  - Pfizer Investigational Site, Tlalpan, Mexico DF
- Pfizer Investigational Site, Amsterdam, North Holland, Netherlands
- Poland (3):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Wroclaw
- Slovakia (3):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Nitra
- South Africa (5):
  - Pfizer Investigational Site, Overport, Durban
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Claremont, Western Cape
  - Pfizer Investigational Site, Durbanville, Western Cape
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Majadahonda, Madrid
- Sweden (2):
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Vaxjo
- United Kingdom (3):
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Lichtenstein GR, Bressler B, Francisconi C, Vermeire S, Lawendy N, Salese L, Sawyerr G, Shi H, Su C, Judd DT, Jones T, Loftus EV. Assessment of Safety and Efficacy of Tofacitinib, Stratified by Age, in Patients from the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):27-41. doi: 10.1093/ibd/izac084. PMID 36342120
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Loftus EV, Baumgart DC, Gecse K, Kinnucan JA, Connelly SB, Salese L, Su C, Kwok KK, Woolcott JC, Armuzzi A. Clostridium difficile Infection in Patients with Ulcerative Colitis Treated with Tofacitinib in the Ulcerative Colitis Program. Inflamm Bowel Dis. 2023 May 2;29(5):744-751. doi: 10.1093/ibd/izac139. PMID 35792493
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- [Derived] Mukherjee A, Tsuchiwata S, Nicholas T, Cook JA, Modesto I, Su C, D'Haens GR, Sandborn WJ. Exposure-Response Characterization of Tofacitinib Efficacy in Moderate to Severe Ulcerative Colitis: Results From Phase II and Phase III Induction and Maintenance Studies. Clin Pharmacol Ther. 2022 Jul;112(1):90-100. doi: 10.1002/cpt.2601. Epub 2022 Apr 27. PMID 35380740
- [Derived] Dubinsky MC, Magro F, Steinwurz F, Hudesman DP, Kinnucan JA, Ungaro RC, Neurath MF, Kulisek N, Paulissen J, Su C, Ponce de Leon D, Regueiro M. Association of C-reactive Protein and Partial Mayo Score With Response to Tofacitinib Induction Therapy: Results From the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):51-61. doi: 10.1093/ibd/izac061. PMID 35380664
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Sharara AI, Su C, Modesto I, Mundayat R, Gunay LM, Salese L, Sands BE. Efficacy and Safety of Tofacitinib in Ulcerative Colitis Based on Prior Tumor Necrosis Factor Inhibitor Failure Status. Clin Gastroenterol Hepatol. 2022 Mar;20(3):591-601.e8. doi: 10.1016/j.cgh.2021.02.043. Epub 2021 Mar 6. PMID 33684552
- [Derived] Vong C, Martin SW, Deng C, Xie R, Ito K, Su C, Sandborn WJ, Mukherjee A. Population Pharmacokinetics of Tofacitinib in Patients With Moderate to Severe Ulcerative Colitis. Clin Pharmacol Drug Dev. 2021 Mar;10(3):229-240. doi: 10.1002/cpdd.899. Epub 2021 Jan 29. PMID 33513294
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Quirk D, Wang W, Nduaka CI, Mukherjee A, Su C, Sands BE. Efficacy and Safety of Extended Induction With Tofacitinib for the Treatment of Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1821-1830.e3. doi: 10.1016/j.cgh.2020.10.038. Epub 2020 Oct 27. PMID 33127596
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Derived] Sands BE, Taub PR, Armuzzi A, Friedman GS, Moscariello M, Lawendy N, Pedersen RD, Chan G, Nduaka CI, Quirk D, Salese L, Su C, Feagan BG. Tofacitinib Treatment Is Associated With Modest and Reversible Increases in Serum Lipids in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jan;18(1):123-132.e3. doi: 10.1016/j.cgh.2019.04.059. Epub 2019 May 8. PMID 31077827
- [Derived] Sandborn WJ, Panes J, D'Haens GR, Sands BE, Su C, Moscariello M, Jones T, Pedersen R, Friedman GS, Lawendy N, Chan G. Safety of Tofacitinib for Treatment of Ulcerative Colitis, Based on 4.4 Years of Data From Global Clinical Trials. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1541-1550. doi: 10.1016/j.cgh.2018.11.035. Epub 2018 Nov 23. PMID 30476584
- [Derived] Winthrop KL, Melmed GY, Vermeire S, Long MD, Chan G, Pedersen RD, Lawendy N, Thorpe AJ, Nduaka CI, Su C. Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2018 Sep 15;24(10):2258-2265. doi: 10.1093/ibd/izy131. PMID 29850873
- [Derived] Sandborn WJ, Panes J, Zhang H, Yu D, Niezychowski W, Su C. Correlation Between Concentrations of Fecal Calprotectin and Outcomes of Patients With Ulcerative Colitis in a Phase 2 Trial. Gastroenterology. 2016 Jan;150(1):96-102. doi: 10.1053/j.gastro.2015.09.001. Epub 2015 Sep 12. PMID 26376350
- [Derived] Panes J, Su C, Bushmakin AG, Cappelleri JC, Mamolo C, Healey P. Randomized trial of tofacitinib in active ulcerative colitis: analysis of efficacy based on patient-reported outcomes. BMC Gastroenterol. 2015 Feb 5;15:14. doi: 10.1186/s12876-015-0239-9. PMID 25651782
- [Derived] Sandborn WJ, Ghosh S, Panes J, Vranic I, Su C, Rousell S, Niezychowski W; Study A3921063 Investigators. Tofacitinib, an oral Janus kinase inhibitor, in active ulcerative colitis. N Engl J Med. 2012 Aug 16;367(7):616-24. doi: 10.1056/NEJMoa1112168. PMID 22894574
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921063&StudyName=A%20Study%20To%20Investigate%20The%20Safety%20And%20Efficacy%20Of%20%20CP-%20690%2C550%20In%20Patients%20With%20Moderate%20And%20Severe%20Ulcerative%20Colitis.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet matched to CP-690,550 orally twice daily for 8 weeks.
- CP-690,550 0.5 mg: CP-690,550 tablets equivalent to CP-690,550 0.5 milligram (mg) orally twice daily for 8 weeks.
- CP-690,550 3 mg: CP-690,550 tablets equivalent to CP-690,550 3 mg orally twice daily for 8 weeks.
- CP-690,550 10 mg: CP-690,550 tablets equivalent to CP-690,550 10 mg orally twice daily for 8 weeks.
- CP-690,550 15 mg: CP-690,550 tablets equivalent to CP-690,550 15 mg orally twice daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Started | 49 | 31 | 33 | 33 | 49
Treated | 48 | 31 | 33 | 33 | 49
Completed | 35 | 20 | 26 | 31 | 45
Not Completed | 14 | 11 | 7 | 2 | 4
Not completed — Adverse Event | 3 | 2 | 0 | 0 | 2
Not completed — Lack of Efficacy | 5 | 6 | 5 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0 | 1
Not completed — Randomized, not treated | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 0.5 mg: CP-690,550 tablets equivalent to CP-690,550 0.5 mg orally twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg | Total
Number analyzed (Participants) | 49 | 31 | 33 | 33 | 49 | 195
Age, Customized [Number; unit: participants]
  18 to 44 years | 28 | 16 | 18 | 17 | 31 | 110
  45 to 64 years | 16 | 14 | 13 | 15 | 16 | 74
  Greater than or equal to (>=) 65 years | 5 | 1 | 2 | 1 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 14 | 12 | 23 | 89
  Male | 23 | 17 | 19 | 21 | 26 | 106

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response
Description: Clinical response was defined as a decrease from baseline in Mayo score of at least 3 points and at least 30 percent, with accompanying decrease in subscore for rectal bleeding of at least 1 point or absolute subscore for rectal bleeding of 0 or 1. Mayo score: instrument designed to measure disease activity of ulcerative colitis. Total score range: 0 to 12; higher score=more severe disease. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy and physician global assessment, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 8
Population: Full analysis set (FAS): all participants who withdrew as treatment failure (TF) or completed >=1 week dosing, had >=1 valid Mayo score during active double-blind phase. Participants who withdrew as TF=non-responders. Missing data due to reason other than TF were excluded. N (number of participants analyzed)=evaluable participants for the measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 40 | 27 | 31 | 30 | 45
percentage of participants | 47.5 | 29.6 | 51.6 | 63.3 | 80.0

2. Secondary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical remission was defined as a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point. Mayo score:instrument designed to measure disease activity of ulcerative colitis. Total score range: 0 to 12; higher score=more severe disease. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy and physician global assessment, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 8
Population: FAS: all participants who either withdrew as treatment failure TF or completed >=1 week dosing, had >=1 valid Mayo score during active double-blind phase. Participants who withdrew as TF were treated as non-responders. Missing data due to reason other than TF were excluded. N=evaluable participants for the measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 41 | 27 | 31 | 30 | 45
percentage of participants | 12.2 | 7.4 | 35.5 | 50.0 | 42.2

3. Secondary Outcome: Percentage of Participants With Endoscopic Response
Description: Endoscopic response was defined as decrease from baseline in the findings of the flexible proctosigmoidoscopy subscore of the Mayo score at least 1 point. Mayo score: instrument designed to measure disease activity of ulcerative colitis. Total score range: 0 to 12; higher score=more severe disease. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy and physician global assessment, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 40 | 27 | 31 | 30 | 45
percentage of participants | 55.0 | 51.9 | 61.3 | 70.0 | 82.2

4. Secondary Outcome: Percentage of Participants With Endoscopic Remission
Description: Endoscopic remission was defined as the findings of flexible proctosigmoidoscopy subscore of the Mayo score equals 0. Mayo score: instrument designed to measure disease activity of ulcerative colitis. Total score range: 0 to 12; higher score=more severe disease. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy and physician global assessment, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 41 | 27 | 31 | 30 | 45
percentage of participants | 2.4 | 7.4 | 19.4 | 30.0 | 26.7

5. Secondary Outcome: Change From Baseline in Partial Mayo Score at Week 2, 4, 8 and 12
Description: Partial Mayo score was ranged from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores: stool frequency, rectal bleeding and physician's global assessment, each ranged from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe).
Time Frame: Baseline, Week 2, 4, 8, 12
Population: FAS: all participants who either withdrew as TF or completed >=1 week of dosing, had >=1 valid Mayo score during active double-blind phase. Baseline-observation-carried-forward (BOCF) was used for participants who withdrew as TF. Missing data due to reasons other than treatment failure were excluded. N=evaluable participants for the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 46 | 31 | 33 | 33 | 49
units on a scale
  Baseline (n=46, 31, 33, 33, 49) | 5.74 (1.39) | 6.10 (1.35) | 5.82 (1.40) | 5.55 (1.48) | 5.53 (1.19)
  Change at Week 2 (n=41, 31, 29, 28, 47) | -0.63 (1.39) | -1.06 (1.46) | -1.66 (2.18) | -2.11 (2.23) | -2.19 (1.94)
  Change at Week 4 (n=42, 28, 30, 29, 48) | -1.26 (1.67) | -1.32 (1.76) | -2.17 (2.68) | -2.62 (2.14) | -2.75 (2.09)
  Change at Week 8 (n=41, 28, 32, 31, 46) | -1.59 (1.53) | -1.46 (2.01) | -2.50 (2.38) | -2.77 (2.45) | -3.28 (2.02)
  Change at Week 12 (n=38, 27, 30, 29, 45) | -2.26 (2.15) | -1.56 (2.24) | -2.60 (2.44) | -3.03 (2.08) | -3.22 (2.31)

6. Secondary Outcome: Change From Baseline in Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 8
Description: IBDQ: Psychometrically validated patient reported outcome (PRO) instrument for measuring disease-specific quality of life (QOL) in participants with IBD. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is sum of each item score, ranged from 32 to 224 with higher score indicates better QOL. Positive change in total score indicated improvement in QOL.
Time Frame: Baseline, Week 8
Population: FAS: all participants who either withdrew as TF or completed >=1 week of dosing, had >=1 valid Mayo score during active double-blind phase. Missing data were excluded. N=evaluable participants for the measure. n=number of participants at specified time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 47 | 31 | 30 | 31 | 48
units on a scale
  Baseline (n=47, 31, 30, 31, 48) | 123.15 (29.46) | 123.81 (34.48) | 132.30 (33.57) | 134.46 (32.50) | 123.95 (34.86)
  Change at Week 8 (n=34, 18, 24, 26, 42) | 27.75 (29.75) | 27.72 (33.37) | 30.29 (27.29) | 30.38 (39.76) | 50.71 (35.55)

7. Secondary Outcome: Change From Baseline in Level of C-Reactive Protein (CRP) at Week 4 and 8
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 4, 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 48 | 31 | 33 | 32 | 49
milligram per liter (mg/L)
  Baseline (n=48, 31, 33, 32, 49) | 9.70 (12.84) | 18.80 (29.43) | 12.55 (13.21) | 11.32 (16.45) | 17.14 (26.44)
  Change at Week 4 (n=38, 22, 25, 30, 46) | -0.70 (6.75) | -4.11 (27.08) | -1.88 (12.41) | -5.68 (13.09) | -9.08 (15.44)
  Change at Week 8 (n=37, 21, 27, 28, 44) | 0.90 (16.41) | -6.84 (27.32) | -3.85 (8.74) | -0.12 (31.33) | -8.20 (21.86)

8. Secondary Outcome: Change From Baseline in Level of Fecal Calprotectin at Week 2, 4, 8 and 12
Description: Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligram per kilogram (mg/kg)
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 46 | 29 | 31 | 32 | 49
milligram per kilogram (mg/kg)
  Baseline (n=46, 29, 31, 32, 49) | 1733 (2596) | 1440 (1623) | 1474 (2182) | 1145 (2001) | 1523 (2575)
  Change at Week 2 (n=39, 24, 28, 31, 47) | -225 (2990) | 1465 (5399) | -65 (3823) | -127 (2212) | -598 (2378)
  Change at Week 4 (n=37, 22, 27, 28, 45) | -512 (2602) | -401 (1789) | -369 (3211) | -681 (1981) | -687 (1941)
  Change at Week 8 (n=40, 25, 28, 31, 43) | -400 (2814) | -292 (1650) | -570 (1797) | -636 (2221) | -596 (4152)
  Change at Week 12 (n=33, 19, 24, 28, 42) | -791 (2290) | 565.7 (2808) | -414 (2245) | -721 (2099) | -753 (1917)

9. Secondary Outcome: Plasma Concentration of CP-690,550
Description: Summary statistics were calculated for each dose group using the nominal collection times and by setting concentration values below the lower limit of quantification (LLOQ) (LLOQ=0.1 nanogram per milliliter [ng/mL]) to zero.
Time Frame: 0.25, 0.5, 1, 2 hours post-dose on Day 1, 0 (pre-dose) and 1 hour post-dose on Week 2, Week 4, 0 (pre-dose), 0.25, 0.5, 1, 2 hours post-dose on Week 8
Population: Analysis population included all participants who had at least 1 plasma concentration. N=evaluable participants for this measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Number analyzed (Participants) | 31 | 32 | 33 | 48
ng/mL
  Day 1: 0.25 hours | 1.27 (1.91) | 13.3 (18.4) | 45.5 (53.8) | 44.5 (48.3)
  Day 1: 0.5 hours | 3.5 (2.45) | 23.1 (15.2) | 70.1 (51.5) | 122.0 (80.3)
  Day 1: 1 hour | 4.34 (1.88) | 27.6 (11.6) | 87.1 (38.7) | 131.0 (54.4)
  Day 1: 2 hours | 3.82 (1.58) | 19.5 (7.72) | 62.6 (27.8) | 96.9 (30.8)
  Week 2: 0 hours | 2.16 (2.19) | 11.3 (14.5) | 39.9 (34.7) | 35.4 (50.2)
  Week 2: 1 hour | 3.37 (3.0) | 21.3 (14.1) | 64.8 (41.4) | 102.0 (60.1)
  Week 4: 0 hours | 2.28 (2.61) | 31.1 (110.0) | 26.4 (32.9) | 40.5 (61.4)
  Week 4: 1 hour | 3.4 (2.45) | 23.5 (18.2) | 75.9 (55.3) | 109.0 (57.6)
  Week 8: 0 hours | 0.59 (0.864) | 3.74 (7.19) | 15.9 (31.5) | 12.3 (13.0)
  Week 8: 0.25 hours | 1.6 (1.85) | 11.9 (14.2) | 50.1 (54.1) | 51.8 (64.4)
  Week 8: 0.5 hours | 4.07 (2.69) | 20.3 (12.7) | 78.8 (61.8) | 99.5 (88.1)
  Week 8: 1 hour | 4.41 (2.51) | 25.4 (10.8) | 78.4 (51.9) | 110.0 (62.3)
  Week 8: 2 hours | 6.48 (15.0) | 19.6 (10.1) | 60.6 (35.2) | 92.0 (50.1)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | CP-690,550 0.5 mg | CP-690,550 3 mg | CP-690,550 10 mg | CP-690,550 15 mg
Serious Adverse Events (participants affected / at risk) | 4/48 | 1/31 | 1/33 | 2/33 | 2/49
Other Adverse Events (participants affected / at risk) | 21/48 | 19/31 | 10/33 | 13/33 | 20/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | CP-690,550 0.5 mg (N=31) | CP-690,550 3 mg (N=33) | CP-690,550 10 mg (N=33) | CP-690,550 15 mg (N=49)
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 2
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | CP-690,550 0.5 mg (N=31) | CP-690,550 3 mg (N=33) | CP-690,550 10 mg (N=33) | CP-690,550 15 mg (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 6 | 5 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip exfoliation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1 | 2
Headache (Nervous system disorders) | 2 | 2 | 3 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Pharmacokinetic (PK) parameters and their correlation with clinical response and inflammatory biomarkers were not reported as data from future studies were to be pooled for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.